CLINICAL TRIAL: NCT03100097
Title: A Prospective, Multicenter, Randomized Control Study To Determine Clinical Effectiveness, Patient Wellness and Cost of Pain Related Care of In-Elastic Lumbar Sacral Orthoses Versus Standard Medical Treatment in Patients Presenting With Acute Low Back Pain In Primary Care Centers
Brief Title: A Prospective, Multicenter, Randomized Control Study To Determine Clinical Effectiveness, Patient Wellness and Cost of Pain Related Care of In-Elastic Lumbar Sacral Orthoses Versus Standard Medical Treatment in Patients Presenting With Acute Low Back Pain In Primary Care Centers (The ARREST Study)
Acronym: ARREST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties recruiting patients
Sponsor: Aspen Medical Products (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPR-ORTHO02-2013
Record Dates: First submitted 2017-02-28; First posted 2017-04-04 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Back Pain; Low Back Pain
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Aspen Horizon 627 LSO) (Experimental): Patients receive a lumbar brace, Aspen Horizon 627 LSO, in addition to normal medical management
  Interventions: Device: Aspen Horizon 627 LSO
- Medical Management (No Intervention): Normal medical management

INTERVENTIONS:
Device: Aspen Horizon 627 LSO
  Arms: Intervention (Aspen Horizon 627 LSO)

SUMMARY:
The objective of this study is to evaluate sixty male and non-pregnant female patients diagnosed with acute moderate to severe low back pain with the onset of symptoms within 30 days. To evaluate functional improvement following a 4-week use of an in-elastic lumbar sacral orthosis (LSO) as a treatment modality for acute low back pain.

DETAILED DESCRIPTION:
The objective of this study is to evaluate sixty male and non-pregnant female patients diagnosed with acute moderate to severe low back pain with the onset of symptoms within 30 days. To evaluate functional improvement following a 4-week use of an in-elastic lumbar sacral orthosis (LSO) as a treatment modality for acute low back pain.

ELIGIBILITY:
* Inclusion Criteria:

  o Moderate to complete disability (baseline ODI score of 21 to 80 percent)
* Exclusion Criteria:

  * Pregnant patients
  * Patients considering pregnancy
  * Patients in any other investigational device or drug study
  * Patients unwilling to return for follow up
  * Patients unwilling to provide access to medical claims associated with pain management.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
40% change in Oswestry Disability Index | 4 weeks
  Oswestry Disability Index

SECONDARY OUTCOMES:
Change in Opioid utilization | 4 weeks, 8 weeks, 12 weeks
  Change in Opioid utilization
Number of participants with treatment-related adverse events as assessed by questionnaire | 4 weeks, 8 weeks, 12 weeks
  Were any complications associated wearing of the brace noted in patients questionnaires
General Health Survey | 12 weeks
  SF36v2 Health Survey